CLINICAL TRIAL: NCT06261138
Title: Survival Analysis of TACE Monotherapy vs. Combination Therapy in BCLC B and C Stage Hepatocellular Carcinoma: A Retrospective Cohort Study
Brief Title: Survival Analysis: TACE vs. Combination Therapy in HCC
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Clinical Professor, Zhejiang University
Other Study IDs: RSR-HCC-2019-001
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Transarterial chemoembolization; Combination therapy; Survival
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TACE group: Patients included in the study underwent either conventional TACE (cTACE) or drug-eluting beads TACE (DEB-TACE) procedures performed by experienced interventional radiologists, taking into account tumor burden, patient tolerance, and individual preferences.
  Interventions: Drug: Transarterial chemoembolization
- Combination group: Systemic treatment commenced within one month after the initial TACE procedure, depending on the proper liver function. Anti-angiogenic agents involved in this study mainly comprised multikinase tyrosine kinase inhibitors. ICIs included therapies targeting programmed cell death protein 1 and its ligands.
  Interventions: Drug: Transarterial chemoembolization; Other: Systemic treatment

INTERVENTIONS:
Drug: Transarterial chemoembolization — A 5-French RH catheter was then introduced to the celiac artery, superior mesenteric and artery common hepatic artery for angiography to determine tumor location, quantity, size, and vascularity. After confirmation by C-arm cone-beam computed tomography (CBCT), chemoembolization was administered by superselective catheterization of the branches of the tumor-feeding arteries using a 2.8-French coaxial microcatheter. For cTACE, oxaliplatin, raltitrexed and an emulsion containing idarubicin and ethiodized oil were infused for over 20 minutes, followed by combined embolization with blank embolic microspheres. For DEB-TACE, DC/LC Beads® (Biocompatibles, Farnham, Surrey, UK), as drug carriers and embolic materials, were loaded with doxorubicin hydrochloride and mixed with nonionic contrast medium. Real-time assessment of embolization was performed with the assistance of CBCT.
  Other Names: TACE
Other: Systemic treatment — sorafenib (Bayer HealthCare, Berlin, Germany), lenvatinib (Eisai, Tokyo, Japan), apatinib (Hengrui Pharmaceuticals, Lianyungang, China) and donafenib (Zelgen Biopharmaceuticals, Suzhou, China), while a minority of patients received bevacizumab (Innovent Biologics, Suzhou, China).
  sintilimab (Innovent Biologics, Suzhou, China), toripalimab (Junshi Biosciences, Suzhou, China), camrelizumab (Hengrui Pharmaceuticals, Lianyungang, China), tislelizumab (BeiGene, Shanghai, China), pembrolizumab (Merck Sharp & Dohme, NewJersey, USA), nivolumab (Bristol Myers Squibb, New York, USA), atezolizumab (Roche, Basel, Switzerland) and envafolimab (Alphamab Biopharmaceuticals, Suzhou, China).
  Groups: Combination group

SUMMARY:
This retrospective observational study aimed to assess potential improvements associated with systemic therapies in patients receiving transarterial chemoembolization (TACE) for initially unresectable HCC.

DETAILED DESCRIPTION:
Standard treatments provide limited benefits for patients with intermediate or advanced hepatocellular carcinoma (HCC). Recently, recommendations on multimodal treatment regimens for patients with locally advanced HCC have attracted much attention. Therefore, this retrospective research was designed to evaluate the clinical outcomes of TACE alone or in combination with immune and targeted therapy in the primary treatment for patients with intermediate to advanced stage HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes, aged 18-75 years old; (2) HCC was clinically or pathologically diagnosed according to the American Association for Liver Diseases (ASSLD) criteria; (3) One or more tumor lesions could be measured according to modified response evaluation criteria in solid tumors (mRECIST) on enhanced CT or MRI; (4) For patients with Barcelona Clinic Liver Cancer (BCLC) stage B or stage C hepatocellular carcinoma (HCC) in Barcelona, and who are not suitable for surgical resection, it is recommended to undergo transarterial chemoembolization (TACE) or combination therapy involving TACE as the initial treatment; (5)Child-Pugh grade A or B, no hydrothorax, ascites and hepatic encephalopathy requiring treatment; (6) Eastern Cooperative Oncology Group performance status (ECOG-PS) score 0-1; (7) Have enough liver and kidney function in patients with appropriate laboratory indicators: hemoglobin concentration (HGB) hemoglobin, acuity 9.0 g/dl, neutrophils acuity 1500 cells/mm3, PLT 50 * 109 / L, or serum propagated 28 g/L, or TBIL< 50umol/L, ALT, AST< 5 times the upper limit of normal, Bun, Cr< 1.5 times the upper limit of normal, INR< 1.7 or PT prolongation < 4s

Exclusion Criteria:

1. Other malignant tumors outside HCC, such as liver metastasis of colon cancer; (2) Child-Pugh grade C; (3) Contraindications to TACE, lenvatinib or tislelizumab; (4) Any active autoimmune diseases or autoimmune disease, thyroid function hyperfunction or decline, which is to be bronchodilator treatment of asthma; (5) There are serious complications, including serious heart, lung, kidney, blood coagulation dysfunction; Important cardiovascular diseases such as heart disease of the definition of New York heart association level 3 or higher, instability during the treatment of myocardial infarction, arrhythmia, unstable angina, etc; (6) Past history of patients with idiopathic pulmonary fibrosis , Machine pneumonia (e.g., occlusive bronchiolitis), drug pneumonia, idiopathic pneumonia or chest CT screening to find evidence for an active pneumonia; (7) Patients with previous allogeneic stem cell or solid organ transplantation, including patients after liver transplantation; (8) Clinical data absence or incomplete information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with treatment-naive intermediate or advanced HCC who received with TACE alone or the combination therapy (TACE plus antiangiogenic agents with or without ICIs) at our institution
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per mRECIST | 12-48 months
  The duration from treatment initiation to PD in patients who cannot undergo surgery, or to the date of postoperative relapse in patients who receive surgery, or death for any reason, whichever occurs first (according to mRECIST).

SECONDARY OUTCOMES:
12 months PFS rate | 12 months
  The percentage of patients who have not progressed or relapsed or death at the 12 month time point since the first time of treatment.
Overall survival (OS) | 24-48 months
  The duration from treatment initiation to death from any cause.
Objective Response Rate (ORR) per mRECIST | 12-48 months
  The proportion of complete response or partial response as optimal response among all treated patients according to mRECIST.
Disease Control Rate (DCR) per mRECIST | 12-48 months
  The proportion of complete response, partial response or stable disease as optimal response among all treated patients according to mRECIST.
Adverse events (AEs) | 12-48 months
  The incidence, relationship with study drugs, and severity level of all adverse events (AEs) according to CTCAE 5.0, treatment-emergent adverse events (TEAEs), treatment related adverse events (TRAEs), and serious adverse events (SAEs) and the changes in vital signs, physical examination results, and laboratory test results before, during, and after the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No